CLINICAL TRIAL: NCT01705730
Title: Mon-ACT: A Multi-center, Non-interventional Study in Rheumatoid Arthritis (RA) Patients Treated With Tocilizumab in Monotherapy
Brief Title: A Non-Interventional Study of Rheumatoid Arthritis Patients Treated With RoActemra/Actemra (Tocilizumab) in Monotherapy
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28269
Record Dates: First submitted 2012-10-10; First posted 2012-10-12 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Tocilizumab: Participants with rheumatoid arthritis (RA) received tocilizumab monotherapy according to individualized physician-prescribed regimens.
  Interventions: Drug: tocilizumab

INTERVENTIONS:
Drug: tocilizumab — Participants received tocilizumab monotherapy according to individualized physician-prescribed regimens.
  Other Names: Actemra

SUMMARY:
This observational study will evaluate the use and efficacy of RoActemra/Actemra (tocilizumab) in monotherapy in routine clinical practice in participants with rheumatoid arthritis. Eligible participants initiated on RoActemra/Actemra treatment according to the licensed label will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Moderate to severe rheumatoid arthritis according to the revised (1987) ACR criteria
* Participants in whom the treating physician has made the decision to commence RoActemra/Actemra treatment in monotherapy in accordance with the local label and the reimbursement criteria indicating that RoActemra/Actemra can be given in monotherapy in case of methotrexate intolerance or where continued treatment with methotrexate is inappropriate; this can include participants who have received RoActemra/Actemra treatment within 8 weeks prior to the enrolment visit
* Concomitant treatment with NSAIDs and/or corticosteroids is allowed

Exclusion Criteria:

* Participants who have received RoActemra/Actemra more than 8 weeks prior to the enrolment visit
* Participants who have previously received RoActemra/Actemra in a clinical trial or for compassionate use
* Participants receiving concomitant DMARD treatment for rheumatoid arthritis at baseline (e.g. hydroxychloroquine, sulfasalazine, methotrexate, leflunomide, gold compounds, cyclosporine) will be excluded from the study
* Participants who have received treatment with an investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever is longer) before starting treatment with RoActemra/Actemra
* Participants with a history of autoimmune disease or any joint inflammatory disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with rheumatoid arthritis initiating treatment with RoActemra/Actemra in monotherapy
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2012-07-31 (Actual); Primary Completion 2014-12-12 (Actual); Study Completion 2014-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- Belgium (17):
  - ASZ Aalst, Aalst
  - CH EpiCURA Site Ath, Ath
  - CHU Brugmann (Victor Horta), Brussels
  - Hospital Erasme; Neurologie, Brussels
  - Reumaclinic, Genk
  - GHdC Site Saint-Joseph, Gilly (Charleroi)
  - Clinique Notre Dame de Grâce, Gosselies
  - CH Jolimont - Lobbes (Jolimont), Haine-Saint-Paul
  - AZ Groeninge, Kortrijk
  - Chr de La Citadelle, Liège
  - Clinique Saint-Joseph, Liège
  - CHU Ambroise Paré, Mons
  - AZ Damiaan, Ostend
  - Clinique St Pierre asbl, Ottignies
  - AZ Delta (Campus Wilgenstraat), Roeselare
  - AZ Turnhout Sint Jozef, Turnhout
  - Sint Augustinus Wilrijk, Wilrijk

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 71 participants were enrolled in the study. Out of 71 participants, 68 received at least one dose of tocilizumab during the study and were included in the full analysis set.
Groups:
- Tocilizumab: Participants with RA received tocilizumab monotherapy according to individualized physician-prescribed regimens.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 68 (Participants who received study drug)
Completed | 59
Not Completed | 9
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1
Not completed — Reason not Specified | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on Tocilizumab Treatment at Month 6 After Treatment Initiation
Time Frame: Month 6 after treatment initiation
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
percentage of participants | 79.4 [67.9 to 88.3]

2. Secondary Outcome: Percentage of Participants With Systemic Manifestations of RA at Baseline
Description: Systemic manifestations of RA included anemia, fatigue, conventional risk factors for cardiovascular disease, C-Reactive Protein (CRP) above upper limit of normal, rheumatoid nodules, rheumatoid vasculitis and interstitial lung disease. Participants were included if they experienced at least any one of the conditions.
Time Frame: Baseline
Population: Data for this outcome measure was not collected.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Disease-Modifying Antirheumatic Drugs (DMARDs) Intolerance and Inadequate Response
Time Frame: Baseline
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
participants
  DMARD Intolerance | 1
  Inadequate Response | 67

4. Secondary Outcome: Number of Participants With Inadequate Response to Other Biologics
Time Frame: Baseline
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
participants | 35

5. Secondary Outcome: Time to Addition of Disease-Modifying Anti-rheumatic Drugs (DMARDs)
Description: The time to DMARD addition equals to the time (days) between tocilizumab start and first start date of DMARDs.
Time Frame: Month 6
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study. Here, number of participants analyzed are the participants who had addition of DMARDs during study.
Measure: Median (Full Range); unit: days
Arm/Group | Tocilizumab
Number analyzed (Participants) | 1
days | 84 [84 to 84]

6. Secondary Outcome: Percentage of Participants Who Had DMARDs During Study
Time Frame: Month 6
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study. Here, number of participants analyzed signifies those participants who had addition of DMARDs during study.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 1
percentage of participants
  Hydroxychoroquine | 0.0
  Sulfasalazine | 0.0
  Methotrexate | 100.0
  Leflunomide | 0.0
  Gold compunds | 0.0
  Cyclosporine | 0.0
  Azatioprine | 0.0
  Other DMARD | 0.0

7. Secondary Outcome: Number of Participants With Dose Reductions
Time Frame: 6 months
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
participants | 4

8. Secondary Outcome: Number of Participants With Starting Tocilizumab After Failing DMARDs
Time Frame: Baseline
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
participants | 33

9. Secondary Outcome: Number of Participants With Starting Tocilizumab After Stopping Other Biologic Agents
Time Frame: Baseline
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
participants | 35

10. Secondary Outcome: Time to Reduction/Withdrawal of Corticosteroids
Time Frame: Month 6
Population: Data was not collected for this outcome measure.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Dose Modifications Per Participant at Month 6
Description: Number of dose modification per participant at Month 6 was reported.
Time Frame: Month 6
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study.
Measure: Mean (Standard Deviation); unit: number of dose modifications
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
number of dose modifications | 0.1 (0.2)

12. Secondary Outcome: Mean Dosing Interval Per Participant at Month 6
Time Frame: Month 6
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study. Analysis was performed only participants reaching 6 month visit.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tocilizumab
Number analyzed (Participants) | 54
days | 25.86 (2.64)

13. Secondary Outcome: Percentage of Participants Discontinued From Tocilizumab for Safety Versus Efficacy
Time Frame: Month 6
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study. Here, number of participants analyzed signifies the participants who were evaluable for the outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 13
percentage of participants
  Adverse Event | 61.5
  Lack of efficacy | 7.7
  Other | 30.8

14. Secondary Outcome: Time for Restoration of Initial Dosing Regimen
Time Frame: Month 6
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study. Here, number of participants analyzed signifies number of participants evaluated for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Tocilizumab
Number analyzed (Participants) | 4
days | NA [NA to NA] — Median and full range could not be reached as less than 50% of the participants restored to initial dosing regimen.

15. Secondary Outcome: Percentage of Participants Who Were Not Adhering to Recommended Dosing Regimen
Time Frame: Month 6
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
percentage of participants | 20.6 [11.7 to 32.1]

16. Secondary Outcome: Number of Participants Who Were Not Adhering to Recommended Management of AEs
Time Frame: Month 6
Population: Only participants experiencing 'adverse events and/or abnormal laboratory tests requiring modification of drug dosage' are taken into account for this analysis.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 8
participants | 0

17. Secondary Outcome: Percentage of Participants Still on Tocilizumab Monotherapy at Month 6
Time Frame: Month 6
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
percentage of participants | 98.1 [90.0 to 99.9]

18. Secondary Outcome: Percentage of Participants With Reason for Choice of Monotherapy at Baseline
Time Frame: Baseline
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
percentage of participants
  MTX Intolerance | 61.8
  Continued MTX not Appropriate | 38.2

19. Secondary Outcome: Tender Joint Count (TJC)
Description: TJC was determined by examining 28 and 68 joints and identifying the joints that were painful under pressure or to passive motion. Tenderness was recorded on the joint assessment form at baseline, no tenderness = 0, tenderness = 1.
Time Frame: Baseline, Month 3, 6
Population: Full analysis set included all participants that received at least one dose of tocilizumab during the study. Here, n signifies the number of participants who were evaluated for the specified time points.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
tender joints
  Baseline for TJC28 (n=47) | 10.3 (6.0)
  Month 3 for TJC28 (n=29) | 2.9 (5.0)
  Month 6 for TJC 28 (n=17) | 2.2 (3.3)
  Baseline for TJC68 (n=7) | 8.6 (3.2)
  Month 3 for TJC68 (n=10) | 2.0 (2.7)
  Month 6 for TJC68 (n=1) | 0.0 (NA) — Standard deviation was not estimable for TJC68 as only 1 participant was evaluated at Month 6.

20. Secondary Outcome: Swollen Joint Count (SJC)
Description: SJC was determined by examining 28 and 66 joints and identifying when swelling was present. Swelling was recorded on the joint assessment form at baseline, no swelling = 0, swelling =1.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
swollen joints
  Baseline for SJC28 (n=47) | 7.9 (5.6)
  Month 3 for SJC28 (n=29) | 1.5 (3.5)
  Month 6 for SJC 28 (n=17) | 0.9 (1.4)
  Baseline for SJC66 (n=7) | 8.9 (4.5)
  Month 3 for SJC66 (n=10) | 0.6 (1.3)
  Month 6 for SJC66 (n=1) | 0.0 (NA) — Standard deviation was not estimable for SJC66 as 1 participant was evaluated at Month 6.

21. Secondary Outcome: Percentage of Participants With Disease Activity Score-28 (DAS28)
Description: DAS28 was calculated from SJC and TJC using 28 joints count, erythrocyte sedimentation rate (ESR) (millimeter per hour [mm/hr]), and patient global assessment of disease activity (PGH) (measured on a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS) where 0=no disease activity and 100=worst disease activity). DAS28 is a measurement of RA activity on a 0 to 10 scale: a score greater than (>) 5.1 indicates high disease activity; a score between 3.2 and 5.1 indicates moderate disease activity; a score of less than 3.2 indicates low disease activity; a score of less than (<) 2.6 is considered remission.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
percentage of participants
  LDA at Baseline (n=38) | 0
  LDA at Month 3 (n=19) | 73.7
  LDA at Month 6 (n=11) | 81.8
  Remission at Baseline (n=38) | 0
  Remission at Month 3 (n=19) | 68.4
  Remission at Month 6 (n=11) | 81.8

22. Secondary Outcome: Percentage of Participants With Good European League Against Rheumatism (EULAR) Response at Month 3 and Month 6
Description: Clinical response assessed as per EULAR categorical DAS28 response criteria was defined as clinically meaningful improvement at a particular time point. EULAR response was based on change from baseline (CFB) in the DAS28 score and also on the actual DAS28 score at the time point so was more reflective of the current status of the participant. EULAR Good response: DAS28 <=3.2 and a CFB <-1.2. EULAR Moderate response: DAS28 >3.2 to ≤ 5.1 or a CFB < -0.6 to ≥ -1.2. EULAR No response: DAS28 ≤3.2 or CFB greater than or equal to (>=) -0.6, DAS28 >3.2 to <=5.1 or CFB>=-0.6 and DAS28 >5.1 or CFB >=-0.6. The DAS28 score was a measure of the participant's disease activity, based on the TJC (28 joints), SJC (28 joints), PGH, and ESR. DAS28 total scores ranged from 0 to approximately 10. Scores <2.6 = best disease control and scores >5.1 = worse disease control. A negative CFB indicated clinically meaningful improvement.
Time Frame: Month 3, 6
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
percentage of participants
  Month 3 (n=10) | 90
  Month 6 (n=5) | 80

23. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) Response at Month 3 and Month 6
Description: ACR response was calculated based on total joint count evaluation (28 or 66/68 joint count) and other clinical and laboratory assessments. A positive ACR20 response required at least a 20% improvement (reduction) compared to baseline in swollen joint count (66 joints) and tender joint count (68 joints) and at least 3 of the following 5 assessments: patient's global assessment of pain, PGH, PhGH (all 3 assessed at 0 [good] to 100 mm [worst] VAS scale), participant assessment of disability measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessed on a 0 to 3 scale, where higher scores represented higher disease activity), Acute phase reactant (CRP or ESR). A reduction in the level of and acute phase reactants was considered an improvement. ACR50, ACR70, ACR90 require a 50%, 70%, 90% improvement from baseline respectively.
Time Frame: Month 3, 6
Population: The ACR analysis was not performed because the Health Assessment Questionnaire (HAQ) disability index score is needed; only HAQ total score expressed in % was available.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

24. Secondary Outcome: Percentage of Participants With Disease Activity According to Clinical Disease Activity Index (CDAI) Response
Description: CDAI is the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PGH and physician global assessment of disease activity (PhGH) assessed on 0-10 cm VAS; 0 = no disease activity and 10 = worst disease activity. CDAI total score = 0-76. CDAI <= 2.8 indicates clinical remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high (or severe) disease activity.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
percentage of participants
  Baseline Remission (n=30) | 0
  Remission at Month 3 (n=8) | 75.0
  Remission at Month 6 (n=4) | 75.0
  Baseline LDA (n=30) | 13.3
  LDA at Month 3 (n=8) | 25.0
  LDA at Month 6 (n=4) | 25.0
  Baseline Moderate Disease Activity (n=30) | 50.0
  Moderate Disease Activity at Month 3 (n=8) | 0
  Moderate Disease Activity at Month 6 (n=4) | 0
  Baseline High Disease Activity (n=30) | 36.7
  High Disease Activity at Month 3 (n=8) | 0
  High Disease Activity at Month 6 (n=4) | 0

25. Secondary Outcome: Percentage of Participants With Disease Activity According to Simplified Disease Activity Index (SDAI) Response
Description: The SDAI was a combined index for measuring disease activity in RA which reflected the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, PGH and PhGH, assessed on 0-100 mm VAS where 0 = no disease activity and 100 = worst disease activity, and C-reactive protein (CRP). SDAI total score = 0-86. A SDAI score </= 3.3 represented clinical remission, a score of between 3.4 and 11.0 represented low disease activity, a score between 11 and 26.0 represented moderate disease activity and a score > 26.0 represented high (or severe) disease.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
percentage of participants
  Baseline Remission (n=28) | 0
  Remission at Month 3 (n=8) | 75.0
  Remission at Month 6 (n=4) | 75.0
  Baseline LDA (n=28) | 17.9
  LDA at Month 3 (n=8) | 25.0
  LDA at Month 6 (n=4) | 25.0
  Baseline Moderate Disease Activity (n=28) | 46.4
  Moderate Disease Activity at Month 3 (n=8) | 0
  Moderate Disease Activity at Month 6 (n=4) | 0
  Baseline High Disease Activity (n=28) | 35.7
  High Disease Activity at Month 3 (n=8) | 0
  High Disease Activity at Month 6 (n=4) | 0

26. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Month 3 and Month 6
Description: The Patient Global Assessment of disease activity provides an overall assessment of how RA affects the participant using a visual analogue score, where 0 indicates they are managing very well and 100 indicates they are managing very poorly. A decrease in the score indicates improvement.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
units on a scale
  Baseline (n=40) | 65.6 (15.2)
  Change at Month 3 (n=12) | -27.8 (27.5)
  Change at Month 6 (n=7) | -30.1 (16.2)

27. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity at Month 3 and Month 6
Description: The physician's global assessment of disease activity was assessed using a 0 to 100 mm horizontal VAS by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
units on a scale
  Baseline (n=34) | 57.6 (23.1)
  Change at Month (n=9) | -41.9 (22.6)
  Change at Month (n=3) | -53.0 (20.7)

28. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) at Month 3 and Month 6
Description: The HAQ was a participant self-reported questionnaire for assessing the extent of a participant's functional ability. It consisted of 20 questions in 8 categories (dressing and grooming, rising, eating, walking, reach, grip, hygiene, and carrying out daily activities). Each question had 4 response options, ranging from 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. The HAQ scale was an average of all the scores and ranged from 0 to 3, where higher scores represented higher disease activity.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
units on a scale
  Baseline (n=42) | 41.11 (19.40)
  Change at Month 3 (n=13) | -23.59 (29.09)
  Change at Month 6 (n=6) | -11.94 (19.87)

29. Secondary Outcome: Change From Baseline in VAS-Fatigue at Month 3 and Month 6
Description: The VAS-fatigue provides an overall assessment of the level of fatigue that the participant is experiencing using a visual analogue score, where 0 indicates no fatigue and 100 indicates extreme fatigue. A decrease in the score indicates improvement.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
units on a scale
  Baseline (n=31) | 64 (16.5)
  Change at Month 3 (n=9) | -19.3 (18.4)
  Change at Month 6 (n=5) | -38.4 (21.4)

30. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Pain at Month 3 and Month 6
Description: The Patient Global Assessment of pain provides an overall assessment of the severity of pain that the participant is experiencing using a visual analogue score, where 0 indicates no pain and 100 indicates unbearable pain. A decrease in the score indicates improvement.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
units on a scale
  Baseline (n=34) | 60.6 (22.9)
  Change at Month 3 (n=9) | -31.8 (25.1)
  Change at Month 6 (n=4) | -33.0 (18.2)

31. Secondary Outcome: Change From Baseline in VAS-Morning Stiffness at Month 3 and Month 6
Description: Morning stiffness was defined by the time elapsed between the time of usual awakening (even if not in the morning) and the time the participant was as limber as he/she would be during a day involving typical activities. Morning stiffness was assessed on a 100 mm VAS, where 0= none and 100= very severe.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
units on a scale
  Baseline (n=22) | 37.8 (22.9)
  Change at Month 3 (n=5) | -7.6 (26.3)
  Change at Month 6 (n=3) | -30.3 (18.5)

32. Secondary Outcome: Percentage of Participants With an Adverse Event (AEs), Serious Adverse Events (SAEs), AEs of Special Interest (AESIs)
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. An Serious Adverse Events (SAEs) is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect. AESI included- serious/medically significant infections; myocardial Infarction/acute coronary syndrome; gastrointestinal perforations; malignancies; anaphylaxis/hypersensitivity reactions; demyelinating disorders; stroke; serious/medically significant bleeding events; serious/medically significant hepatic events.
Time Frame: Month 6
Population: Safety population included all participants that received a dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
percentage of participants
  AE | 61.8
  SAE | 4.4
  AESI | 8.8

33. Secondary Outcome: Percentage of Participants With AEs Leading to Dose Modifications
Time Frame: Month 6
Population: Safety population included all participants that received a dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
percentage of participants | 7.4

34. Secondary Outcome: C-reactive Protein (CRP]) Level
Description: CRP is an acute phase reactant and is a measure of inflammation.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
milligram per liter (mg/L)
  Baseline (n= 51) | 9.94 (20.71)
  Month 3 (n= 52) | 5.04 (18.95)
  Month 6 (n= 28) | 2.49 (3.16)

35. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) Level
Description: ESR is an acute phase reactant and is a measure of inflammation.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: millimeter per hour (mm/hr)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
millimeter per hour (mm/hr)
  Baseline (n= 42) | 24.31 (24.68)
  Month 3 (n= 38) | 12.71 (23.84)
  Month 6 (n= 17) | 8.88 (15.07)

ADVERSE EVENTS:
Time Frame: Month 6
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 3/68
Other Adverse Events (participants affected / at risk) | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=68)
Sarcoidosis (Immune system disorders) | 1
Depression (Psychiatric disorders) | 1
Infarction (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.